CLINICAL TRIAL: NCT06214845
Title: Early-goal Directed Automated Red Blood Cell Exchange for Acute Chest Syndrome in Sickle Cell Disease: a Multicentre, Randomised, Clinical Trial
Brief Title: Early-goal Directed Automated Red Blood Cell Exchange for Acute Chest Syndrome in Sickle Cell Disease
Acronym: ARCAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230784
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Acute Chest Syndrome
Keywords: Sickle cell disease (SCD); Acute chest syndrome (ACS); Red blood cell exchange (REX); Oxygen; Respiratory support
MeSH Terms: conditions — Acute Chest Syndrome; Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: A multicentre, randomised, controlled, superiority clinical trial. Participants will be randomly assigned to one of the two groups of the study (manual or automated REX) with a 1:1 allocation as per a computer generated randomisation list stratified by site and type of respiratory support as follows: low flow-oxygen vs noninvasive respiratory support (i.e., high low oxygen or continuous positive airway pressure or noninvasive ventilation) vs invasive ventilation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated REX (Experimental): Automated REX
  Interventions: Procedure: Red blood cell EXchange (REX)
- Manual REX (Active Comparator): First manual REX will be performed as soon as possible after randomisation, and the patient will be re-assessed every 24 hours (repeated manual REX will be allowed in case of clinical worsening after 24 or 48 hours or in the absence of clinical improvement after 72 hours)
  Interventions: Procedure: Red blood cell EXchange (REX)

INTERVENTIONS:
Procedure: Red blood cell EXchange (REX) — A single automated REX will be performed, as soon as possible after randomization.
  Other Names: Automated REX

SUMMARY:
Sickle cell disease (SCD) is characterized by recurrent vaso-occlusive pain crisis (VOC), which may evolve to acute chest syndrome (ACS), the most common cause of death among adult patients with SCD. Currently, there is no etiologic treatment to abort ACS. Therefore, management of ACS mostly involve a symptomatic approach including in routine, and as per recommendations, hydration, analgesics, supplemental oxygen, and transfusion.

The polymerisation of sickle haemoglobin (HbS) is one major feature in the pathogenesis of vaso-occlusion. Current guidelines recommend red blood cell exchange transfusion (REX) in patients with severe ACS in order to improve oxygenation and reduce HbS concentration to blunt sickling. REX is often preferred over simple transfusion in this setting because it rapidly reduces HbS without raising final haematocrit. There are currently two methods for REX: manual (with sequential phlebotomies and transfusions) or automated (erythrocytapheresis). The former allows a sober use of red blood cell packs, while the latter achieves haematological targets (HbS and haematocrit) quickly and more consistently, but requires a special equipment and trained staff. As a result of inflammation and intravascular hemolysis, the plasma of patients with ACS may also contain several components that promote vaso-occlusion, lung injury and organ failure, including cytokines (e.g., IL-6), free haemoglobin and free haem. Conversely, it is depleted in haptoglobin and hemopexin, which normally bind to and clear cell-free haemoglobin. The addition of therapeutic plasma exchange to erythrocytapheresis during automated REX may therefore have a dual beneficial effect in patients with overt intravascular hemolysis: i) deplete the inflammatory mediators and products of hemolysis; ii) replete haptoglobin and hemopexin. REX modalities (automated vs manual) have not been tested during ACS.

The hypothesis is that early-goal directed automated REX may accelerate the resolution of severe ACS as compared to manual REX.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with major sickle cell disease syndrome (SS, SC, Sβ0 or Sβ+)
* ACS, as defined by the association of fever and/or acute respiratory symptoms with a new pulmonary infiltrate on chest imaging
* Requiring supplemental oxygen ≥ 2 L/min for SpO2 ≥ 95%
* With an indication for REX given the hypoxemic ACS, as per recommendations
* Express informed consent from the relatives or the patient himself, or emergency inclusion procedure in case of inability of patient or proxy relatives to give consent NB: Patients not affiliated to social security will be included in the study given the precarious social situation of many patients with SCD

Exclusion Criteria:

* Patient having both ACS criteria and need for supplemental oxygen ≥ 2 L/min for SpO2 ≥ 95% since more than 72 hours
* Red blood cell transfusion or REX during the current ACS episode
* Any past medical history of delayed haemolytic transfusion reaction
* History of < 12 transfused RBC or anti-red blood cell antibody production on the one hand and no possibility for matching on Rh/K, antibody specificity, and extended to Duffy (Fya), Kidd (Jka and Jkb) and MNS (M, N, S and s) phenotypes on the other hand (12)
* Known legal incapacity (guardianship, curatorship)
* Prisoners or subjects who are involuntarily incarcerated
* Anatomical factors precluding placement of an adequate venous access
* Known pregnancy or current lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of automated (vs manual) REX to reduce time to successful weaning from both supplemental oxygen and any respiratory support (non-invasive or invasive) in adult SCD patients with hypoxemic ACS. | 48 hours after randomization
  Time to successful weaning from both supplemental oxygen and any respiratory support, defined as SpO2 ≥ 95% without oxygen and any respiratory support (non-invasive or invasive) during 48 hours.

SECONDARY OUTCOMES:
Number of participants with complications during hospitalisation and within 3 months following randomisation | Up to 3 months
Time to discharge | Up to 3 months
  Length of hospital stay
Mortality | Up to 3 months
  During hospitalisation and within 28 days and 3 months following randomisation
Number of participants need for noninvasive respiratory support | Up to 28 days
  high flow nasal oxygen, continuous positive airway pressure, or bilevel non-invasive ventilation)
Number of participants readmitted for VOC or ACS | Up to 3 months
Rate of haemoglobin S (HbS) after the first REX and at day-3 | Up to 3 days
Number of participants with change in arterial blood gases and routine biology | 3 and 6 days after randomization
  routine laboratory tests including: complete blood count, arterial blood gas, serum creatinine, aspartate and alanine aminotransferase (AST/ALT), total and direct bilirubin, lactate dehydrogenase (LDH), CRP; blood electrolyte panel
Number of participants with improved chest imaging | 3 and 6 days after randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- Armand MEKONTSO DESSAP, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION